CLINICAL TRIAL: NCT02581566
Title: Effect of Intrathecal vs Intraarticular Dexmedetomidine on Postoperative Pain Following Arthroscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Eman A. Ismail, Lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 01003060215
Record Dates: First submitted 2015-10-18; First posted 2015-10-21 (Estimated); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Intrathecal Dexmedetomidine Group (Active Comparator): 30 patients will be given Intrathecal Dexmedetomidine plus Intrathecal Bupivacaine
  Interventions: Drug: Intrathecal Dexmedetomidine
- Intraarticular Dexmedetomidine Group (Active Comparator): 30 patients will be given Intraarticular Dexmedetomidine plus Intrathecal Bupivacaine
  Interventions: Drug: Intraarticular Dexmedetomidine
- control Group (Other): 30 patients will be given Intrathecal Bupivacaine
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Intrathecal Dexmedetomidine — Addition of Intathecal Dexmedetomidine plus Intrathecal Bupivacaine
  Arms: Intrathecal Dexmedetomidine Group
Drug: Intraarticular Dexmedetomidine — Addition of Intraarticular Dexmedetomidine plus Intrathecal Bupivacaine
  Arms: Intraarticular Dexmedetomidine Group
Drug: Bupivacaine — Intrathecal Bupivacaine
  Arms: control Group

SUMMARY:
Comparison between intrathecal Dexmedetomidine versus Intraarticular Dexmedetomidine on postoperative pain after knee arthroscopy.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, ASA I-II, undergoing knee arthroscopy under spinal anesthesia.

Exclusion Criteria:

* Absolute or relative contraindications to spinal anesthesia, allergy to dexmedetomidine or chronic pain treatment.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2015-07; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
postoperative pain | 24 hours
  Assesment is done by Visual Analog Scale

SECONDARY OUTCOMES:
c-reactive protein | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University Hospital, Asyut, Egypt